CLINICAL TRIAL: NCT06777940
Title: Effects of Kegel Exercises With and Without Myokinetic Active Release of Trigger Points on Pain, Fatigue and Quality of Life in Primary Dysmenorrhea
Brief Title: Effects of Kegel Exercises and Myokinetic Release of Trigger Points in Primary Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Riphah uni
Record Dates: First submitted 2025-01-01; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Primary Dysmenorrhea
Keywords: trigger points

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group A (Experimental): Kegel exercises and Myokinetic active release of trigger points
  Interventions: Other: Kegel exercises

INTERVENTIONS:
Other: Kegel exercises — It consists of 25 patients who will receive Kegel exercises with Myokinetic active release of trigger points in quadratus lumborum, rectus abdominis and gluteus medius. Patient will be in lying position with empty bladder. Ask patient to tight pelvic floor muscle group and hold tight from 3-5 seconds Then relax muscle group from 3-5 seconds with Myokinetic therapy targeted at releasing muscle of quadratus lumborum, rectus abdominis and gluteus medius release was applied passively by sustained pressure for 8-10 seconds. This protocol consisted of three sets with 2 minutes of rest..Participants will be asked to perform exercise 30 times each session following hold and relax of muscle group for 3-5 seconds
  Other Names: myokinetic active release of trigger points; kegel exercise

SUMMARY:
The rationale of this study is despite the widespread belief that exercise can reduce dysmenorrhea, evidence-based studies are limited. Studies are therefore required to evaluate the association between quality of life and the primary dysmenorrheal females, the functional impact on the quality of life and primary dysmenorrhea females also it's a crucial time for females to focus on their studies and dysmenorrhea can add to the fatigue levels and cause distress in this age group thus the purpose of this study is to determine whether myokinetic active release of trigger points in the rectus abdominis, gluteus medius and quadratus lumborum is a more effective way to reduce dysmenorrhea than kegel exercises

DETAILED DESCRIPTION:
Existing research may concentrate on specific interventions or populations, leaving a void in our knowledge of the possible synergistic effects of various exercises when done both alone and in combination, Studies have provided that dysmenorrhea is treated with pelvic floor strengthening however, there is little evidence that myokinetic involvement can lead to progressive outcomes. Given the interdependence of physiology, anatomy and dysfunction. Myokinetic trigger point release may be helpful in promoting the recovery of primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Age 17-25 years
* Diagnosed cases of dysmenorrhea
* Subject having trigger point in rectus abdominins, quadratus lumborum and gluteus medius
* With regular cycles 21-35 days lasting 3-7 days

Exclusion Criteria:

* Oral contraceptives used for menstrual irregularity
* Other gynecological disease like fibroids, endometriosis
* Who take analgesia
* Endometrial polyp, having pelvic infection using IUD, having venous congestion in internal genital organs.

Ages: 17 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Age 17-25 years Diagnosed cases of dysmenorrhea Subject having trigger point in rectus abdominins, quadratus lumborum and gluteus medius With regular cycles 21-35 days lasting 3-7 days
Enrollment: 50 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
pain is assessed by numerical pain rating scale | at baseline pre intervention, at the end of 8 week post intervention
  11 point numeric pain rating scale
FSS scale is used to access fatigue severity | at baseline pre intervention, at the end of 8 week post intervention
  9 items scale
SF-36 is used to access quality of life | at baseline pre intervention, at the end of 8 week post intervention
  8 domains with further items

CONTACTS AND LOCATIONS:
Overall Officials: Iqra abdul ghafoor, PPDPT, Principal Investigator — riphah international univrsity
Locations (2):
- Pakistan (2):
  - Major balqees maternity home, Lahore, Punjab Province
  - Major Balqees Maternity Home Clinic, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Gupta S, Arora M, Yadav PJRJoMS. Comparative Evaluation of Effectiveness of Pelvic Floor Strengthening and Myokinetic Active Release of Trigger Points in Reducing Dysmenorrhea. 2023;13(3) 2. Rani M, Kaushal K, Kaur S. Prevalence of Musculoskeletal Pain and Awareness of Physiotherapy in Primary Dysmenorrhea among Female Students of Adesh University, Bathinda